CLINICAL TRIAL: NCT03381131
Title: The Chinese Version of the Modified American College of Rheumatology (ACR) Diagnostic Criteria for Fibromyalgia and the Fibromyalgia Impact Questionnaire: Reliability and Validity
Brief Title: Chinese Version of Fibromyalgia Criteria and Severity Scales Study
Status: Completed | Type: Observational
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Juan Jiao, Deputy chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: 83376
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Chinese Version; Fibromyalgia; Diagnosis; Fibromyalgia Impact Questionnaire
MeSH Terms: conditions — Fibromyalgia; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Up to now, there is no Chinese version of fibromyalgia diagnosis criteria and severity assessment scales. The aim of this study is to translate, adapt, and validate the Chinese version of the 2011 modification of the 2010 ACR preliminary criteria for the diagnosis of fibromyalgia (2011ModCr) and 2016 ACR revisions to the 2010/2011 fibromyalgia diagnostic criteria, as well as the Fibromyalgia Impact Questionnaire (FIQ-C).

DETAILED DESCRIPTION:
Fibromyalgia is a chronic debilitating musculoskeletal pain syndrome that causes substantial physical and psychological impairments. The provisional criteria of the ACR 2010 and the 2011 self-report modification for survey and clinical research are widely used for fibromyalgia diagnosis. However, there is no Chinese version of fibromyalgia diagnosis criteria and severity assessment scales until now. The aim of this study is to investigate the reliability and the validity of the Chinese version of the 2011ModCr and 2016 ACR revisions to the 2011ModCr, as well as its quantification scale, the Chinese version of Fibromyalgia Impact Questionnaire (FIQ-C) and Revised FIQ (FIQR-C). In this study, we'll divide patients with chronic pain without psychiatric disorders other than depression into two groups according to the 1990 ACR diagnostic criteria for fibromyalgia, a fibromyalgia group and a non-fibromyalgia group. Patients in both groups will be assessed using the 2011ModCr and 2016 ACR revisions to the 2011ModCr. Furthermore, those in the fibromyalgia group will also complete FIQ-C, FIQR-C and several other validated questionnaires including the Medical Outcome Survey Short Form-36 (SF-36), the Beck Depression Inventory (BDI), ect.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Fulfills the American College of Rheumatology (ACR) 1990 classification criteria for Fibromyalgia.

Exclusion Criteria:

* Without any psychiatric disorders other than depression.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The fibromyalgia patients who meet the ACR 1990 criteria for diagnosis without psychiatric disorders other than depression will be recruited. During the study period, other patients with diseases associated with chronic pain, such as rheumatoid arthritis (RA), osteoarthritis (OA), and gout, who have not been diagnosed previously with fibromyalgia will be recruited as control patients. An experienced rheumatologist familiar with fibromyalgia assessed these patients.
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
the Chinese Version of Fibromyalgia Impact Questionnaire (FIQ-C) | up to 1 week
  This questionnaire was designed to assess the current health status of patients with fibromyalgia. The FIQ has 11 individual questions and measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being over the past week ranging from 0-100 with higher score indicating more severity.

SECONDARY OUTCOMES:
Widespread pain index (WPI) | up to 1 week
  WPI is the sum of number of areas (including both jaws, shoulder girdles, upper arms, lower arms, hips (buttocks, trochanters), upper legs and lower legs, as well as neck, shoulder girdle, upper back, lower back, chest and abdomen) in which the patient has had pain over the last week. Its score is between 0 and 19 with higher score indicating more severity.
Symptom severity scale (SSS) | up to 1 week
  The SSS score is the sum of the severity scores of the 3 symptoms (fatigue, waking unrefreshed, and cognitive symptoms) (0-9) plus the sum (0-3) of the number of the 3 symptoms (headaches, pain or cramps in lower abdomen and depression) the patient has been bothered by that occurred during the previous 6 months. Its range is from 0-12 with higher score indicating more severity.
the polysymptomatic distress (PSD) scale | up to 1 week
  The PSD scale fibromyalgia severity (FS) scale also known as the fibromyalgia severity (FS) scale. It is the sum of the WPI and SSS, and ranges is from 0-31 with higher score indicating more severity.
the Chinese Version of the Revised Fibromyalgia Impact Questionnaire (FIQR-C) | up to 1 week
  The FIQR has 21 individual questions and is divided into three linked sets of domains as the FIQ (that is, function, overall impact and symptoms). It differs from the FIQ in having modified function questions and the inclusion of questions on memory, tenderness, balance and environmental sensitivity. The total FIQR is the sum of the three modified domain scores which ranges is also from 0-100 with higher score indicating more sever symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Jiao J, Cheng ZY, Xiao YY, Wang H, Zhang YF, Zhao YY, Jia Y. Validation of the 2011 and 2016 American college of rheumatology diagnostic criteria for fibromyalgia in a Chinese population. Ann Med. 2023;55(2):2249921. doi: 10.1080/07853890.2023.2249921. PMID 37634058
- [Derived] Li YT, Jiang Q, Jia Y, Zhang YF, Xiao YY, Wang H, Zhao YY, Jiao J. A Chinese version of the revised Fibromyalgia Impact Questionnaire: A validation study. Int J Rheum Dis. 2023 Feb;26(2):242-249. doi: 10.1111/1756-185X.14472. Epub 2022 Oct 19. PMID 36261882